CLINICAL TRIAL: NCT00089115
Title: Phase III, Randomized, Double Blind, Placebo-Controlled Trial of Favldand GM-CSF Versus Placebo and GM-CSF Following Rituximab in Subjects With Follicular B-Cell Non-Hodgkin's Lymphoma
Brief Title: Vaccine Therapy and Sargramostim Compared With Placebo and Sargramostim Following Rituximab in Treating Patients With Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn as company has shut down and filed for bankruptcy
Sponsor: Favrille (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: FAV-ID-06; CDR0000378046 (Registry Identifier: PDQ (Physician Data Query)); FAV-WIRB-20040335; CWRU-FVID-1404
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2006-02

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; sargramostim

INTERVENTIONS:
Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine
Biological: rituximab
Biological: sargramostim

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Vaccines made from a person's cancer cells may make the body build an immune response to kill cancer cells. Colony-stimulating factors such as GM-CSF increase the number of immune cells found in bone marrow and peripheral blood. It is not yet known whether combining rituximab and GM-CSF with vaccine therapy may cause a stronger immune response and kill more cancer cells.

PURPOSE: This randomized phase III trial is studying giving rituximab and GM-CSF together with vaccine therapy and comparing it to giving rituximab and GM-CSF alone in treating patients with newly diagnosed, relapsed, or refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare time to disease progression in patients with grade 1, 2, or 3 follicular B-cell non-Hodgkin's lymphoma who respond (i.e., complete or partial response, or stable disease) to treatment with rituximab and are then treated with sargramostim (GM-CSF) with vs without autologous immunoglobulin idiotype-KLH conjugate vaccine.

Secondary

* Compare response rate improvement in patients treated with these regimens.
* Compare overall complete response rate in patients treated with these regimens.
* Compare duration of response in patients treated with these regimens.
* Determine the safety of these regimens in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to prior treatment (yes vs no) and response to rituximab during study (complete response [CR] or partial response [PR] vs stable disease [SD]).

All patients receive rituximab IV once weekly for 4 weeks. Five weeks after the last dose of rituximab, patients are assessed for response. Patients with progressive disease are removed from the study and do not undergo randomization. Patients with a CR, PR, or SD are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive autologous immunoglobulin idiotype-KLH conjugate vaccine subcutaneously (SC) on day 1. Patients also receive sargramostim (GM-CSF) SC on days 1-4.
* Arm II: Patients receive placebo SC on day 1. Patients also receive GM-CSF SC on days 1-4.

In both arms, treatment repeats monthly for 6 months in the absence of unacceptable toxicity or clinically significant progressive disease. After the first 6 months, patients with a CR, PR, or SD may continue to receive treatment (per treatment arm as above) every 2 months for 1 year (total of 6 doses) and then every 3 months thereafter in the absence of disease progression.

Patients are followed every 3 months for 2 years and then every 6 months until disease progression.

PROJECTED ACCRUAL: A total of 342 evaluable patients (171 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular B-cell non-Hodgkin's lymphoma (NHL)

  * Grade 1, 2, or 3
* Meets 1 of the following criteria for treatment with rituximab:

  * Treatment naïve
  * Relapsed or refractory disease after prior chemotherapy
  * Relapsed after a prior documented response (i.e., complete or partial response) to rituximab of at least 6 months duration
* Tumor accessible for biopsy OR existing biopsy material (taken within the past 6 months) suitable for vaccine preparation
* Measurable or evaluable disease after tumor tissue procurement for vaccine production
* No more than 2 prior treatment regimens for NHL

  * Single regimens include any of the following:

    * Maintenance rituximab
    * Rituximab administered once weekly for 8 courses
    * Cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) plus rituximab* NOTE: *CHOP followed by rituximab at time of relapse is considered 2 treatment regimens
* No history of CNS lymphoma or meningeal lymphomatosis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3 (unless related to bone marrow involvement by lymphoma)
* Hemoglobin ≥ 10g/dL

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No congestive heart failure

Pulmonary

* No compromised pulmonary function

Immunologic

* HIV negative
* No prior allergic response to GM-CSF
* No active bacterial, viral, or fungal infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric disorder that would preclude study participation
* No other malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious nonmalignant disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* See Chemotherapy
* At least 4 weeks since prior immunotherapy
* No prior radiolabeled anti-lymphoma antibody (e.g., iodine I 131 tositumomab or ibritumomab tiuxetan)
* No prior autologous or allogeneic stem cell transplantation
* No prior lymphoma-specific idiotype immunotherapy (e.g., Id vaccine)
* No prior investigational vaccine or immunotherapeutic containing keyhole limpet hemocyanin (KLH)

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* More than 9 months since prior fludarabine
* More than 2 years since prior chemotherapy/rituximab combination therapy (e.g., CHOP/rituximab or cyclophosphamide, vincristine, and prednisone [CVP]/rituximab)
* No more than 6 total prior treatment courses with fludarabine

Endocrine therapy

* No concurrent steroids for allergic reaction to sargramostim (GM-CSF)

Radiotherapy

* See Biologic therapy
* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* At least 4 weeks since prior experimental therapy
* No concurrent systemic immunosuppressive therapy
* No other concurrent anti-lymphoma therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-07

PRIMARY OUTCOMES:
Time to progression after 248 patients have progressed

SECONDARY OUTCOMES:
Response rate improvement after 248 patients have progressed
Overall complete response rate by modified Cheson Criteria after 248 patients have progressed
Duration of response by modified Cheson Criteria after 248 patients have progressed
Safety by Common Toxicity Criteria (CTC) after 248 patients have progressed

CONTACTS AND LOCATIONS:
Overall Officials: John F. Bender, PharmD, Study Chair — Favrille
Locations (60):
- United States (60):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Hoag Cancer Center at Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Sharp Memorial Hospital Cancer Center, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Rocky Mountain Cancer Centers - Denver Midtown, Denver, Colorado
  - Medical Oncology Hematology Consultants, P.A. at Helen F. Graham Cancer Center, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Center for Hematology-Oncology - Boca Raton, Boca Raton, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Kaiser Permanente Medical Office - Interstate Medical Office Central, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
  - Baylor University Medical Center - Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Cancer Care Network of South Texas, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin

REFERENCES:
- [Result] Freedman A, Neelapu SS, Nichols C, Robertson MJ, Djulbegovic B, Winter JN, Bender JF, Gold DP, Ghalie RG, Stewart ME, Esquibel V, Hamlin P. Placebo-controlled phase III trial of patient-specific immunotherapy with mitumprotimut-T and granulocyte-macrophage colony-stimulating factor after rituximab in patients with follicular lymphoma. J Clin Oncol. 2009 Jun 20;27(18):3036-43. doi: 10.1200/JCO.2008.19.8903. Epub 2009 May 4. PMID 19414675